CLINICAL TRIAL: NCT00512447
Title: Normal Values of Cerebral Oxygenation
Brief Title: Normal Values of Brain Oxygenation
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Department of Anesthesia, University Hospital Basel
Other Study IDs: EK 62/07
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Cerebral Arterial Disease
Keywords: Aging
MeSH Terms: conditions — Cerebral Arterial Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
New technology allows non-invasive monitoring of brain oxygenation (Near-Infrared-Spectroscopy). However, there are no large series of normal values in various adult age groups. We hypothesised that baseline values in patients breathing room air are lower in old patients than in younger subjects and that younger patients respond increase their brain oxygenation more in response to supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 95 years undergoing a elective surgical procedure

Exclusion Criteria:

* History of cerebral disease
* Dependence on supplemental oxygen

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD, PhD, Principal Investigator — Department of Anaesthesia, University Hospital Basel, Switzerland
Locations (1):
- Department of Anaesthesia, University Hospital Basel, Basel, Canton of Basel-City, Switzerland